CLINICAL TRIAL: NCT01792843
Title: Cognitive Phenotypes in Parkinson's Disease: Anatomical and Functional Correlates
Brief Title: Cognitive Phenotypes in Parkinson's Disease
Acronym: CogPhenoPark
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012_26; 2012-A01317-36. (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease: Patients with Parkinson's disease according to international criteria
  Interventions: Behavioral: data

INTERVENTIONS:
Behavioral: data — * comparisons of clinical characteristics
  * comparisons of cognitive profiles
  * comparisons of grey matter density patterns
  * comparisons of EEG rhythms features

SUMMARY:
* a data driven approach has identified different cognitive phenotypes in Parkinson's disease (PD)
* this heterogeneity possibly reflects the diversity of the neuronal damage caused by the disease
* we hypothesize that the different clinical presentations are associated to specific anatomical and functional correlates

DETAILED DESCRIPTION:
Cognitive impairments are frequent in PD, even in non-demented patients. However, there is a substantial heterogeneity in the clinical presentation of cognitive deficits in PD 2 and also in their progression. This heterogeneity possibly reflects the diversity of the neuronal damage caused by the disease and recent studies suggest that these different clinical influence the risk of developing dementia.

Most studies on cognitive phenotypes in PD have used predefined categories, such as demented vs. non-demented, or PD-mild cognitive impairment vs. cognitively intact patients. However, such an approach may miss less obvious or unexpected presentations. To this end, in a first part of this study, we have used a data-driven approach (cluster analysis) to identify different cognitive phenotypes in PD. With such an approach where phenotypical profiles arise from the data without a priori assumptions, five cognitive presentations were identified: i°) cognitively intact patients (19.39%), ii°) patients with slight mental slowing and mild executive dysfunction (41.29%), iii°) patients with slightly impaired overall cognitive efficiency and deficits in all cognitive domains except recognition memory (12.93%), iv°) patients with severe mental slowing, impaired overall cognitive efficiency, and severe cognitive impairment in all domains, including memory (23.88%), and v°) patients with very severe impairment in all cognitive domains (2.51%). From these results, it could be hypothesized that cognitive deterioration in PD progresses along a continuum, with the exception of the fourth group that also exhibits memory deficits. This group may be characterized by a different underlying pathology, or comorbidity with Alzheimer's disease. The role of vascular factors has also to be considered.

The objectives of the current project are:

1. to validate the identified cognitive profiles prospectively in a new population using confirmatory cluster analysis.
2. to identify specific anatomical correlates for the identified cognitive profiles by magnetic resonance-imaging (MRI) scanning
3. to identify specific functional correlates of the identified cognitive profiles by high-density EEG (hd-EEG)

ELIGIBILITY:
Inclusion Criteria:

* Males or females;
* 18 to 80 years;
* Parkinson's disease, according to international criteria;
* Without neurological co-morbidity;
* Benefiting from health insurance;
* Having read and understood the information form and having signed the consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Parkinsonian syndrome other than PD;
* Currently participating in an other clinical trial or study;
* Patient whose physical or mental condition is incompatible with the study assessments;
* Person under tutorship or curatorship;
* Subjects with claustrophobia
* Subjects carrying incompatible metallic devices such as pacemakers and certain mechanical valves
* PD patients treated by deep brain stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease, according to international criteria, irrespective of their disease stage or their current antiparkinsonian medication
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequency (%) of the cognitive profile | 2 years
  Frequency of the different observed cognitive profile, as coming from the cluster analysis

SECONDARY OUTCOMES:
Grey matter density (voxels) | 2 years
  Grey matter density as measured by voxel-based morphometry

OTHER OUTCOMES:
EEG power (microvolts2) | 2 years
  EEG power in the different frequency bands

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Dujardin, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carey G, Lopes R, Viard R, Betrouni N, Kuchcinski G, Devignes Q, Defebvre L, Leentjens AFG, Dujardin K. Anxiety in Parkinson's disease is associated with changes in the brain fear circuit. Parkinsonism Relat Disord. 2020 Nov;80:89-97. doi: 10.1016/j.parkreldis.2020.09.020. Epub 2020 Sep 19. PMID 32979785